CLINICAL TRIAL: NCT06182384
Title: A Single-center, Randomized, Open, Two-period, Two-sequence Crossover Clinical Study to Compare the Safety and Pharmacokinetics of SHR-1314 Injection in Healthy Subjects at Different Specifications Devices
Brief Title: A Clinical Study to Compare the Safety and Pharmacokinetics of SHR-1314 Injection in Healthy Subjects at Different Specifications Devices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1314-106
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Moderate-to-Severe Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized, open-label, two-period, and two-sequence crossover design trial, consisting of two sequences (sequence A and sequence B) and two periods (first period and second period). Each sequence receives a same dose of SHR-1314 at every period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: SHR-1314
- Sequence B (Experimental)
  Interventions: Drug: SHR-1314

INTERVENTIONS:
Drug: SHR-1314 — Receive a single dose of 240mg SHR-1314 at every period (First period：1mL AI, injection two needles. Second period: 2mL AI, injection one needle).
  Arms: Sequence A
Drug: SHR-1314 — Receive a single dose of 240mg SHR-1314 at every period (First period：2mL AI, injection one needle. Second period: 1mL AI, injection two needles).
  Arms: Sequence B

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of SHR-1314 injection in healthy subjects at different specifications devices.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent form before related activities of the experiment and understanding of the procedures and methods of the experiment, willing to strictly follow the clinical trial protocol to complete the experiment.
2. Both men and women are eligible, aged 18 to 45 years old (inclusive, as determined at the time of signing informed consent form).
3. Body mass index (BMI) is between 18 and 25 kg/m2 (inclusive), with male weight ≥ 50 kg and female weight ≥ 45 kg.
4. Subjects with normal physical examination results and with normal laboratory results (blood, chemistry, urine, drug screening, coagulation function test), ECG and X-ray chest test are normal or with certain abnormal without clinical significance.

Exclusion Criteria:

1. Having a history of any clinically significant disease or condition that the investigator believes may affect the trial results, including but not limited to a history of cardiovascular, endocrine, neurological, digestive, urinary, hematological, immunological, metabolic diseases, or existing diseases in these systems.
2. Have a history of drug or other allergies, or are likely to be allergic to the investigational drug or any component of the investigational drug as determined by the investigator.
3. History or current infection with human immunodeficiency virus (HIV) or hepatitis C; or current hepatitis B infection or syphilis.
4. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years.
5. History of chronic or recurrent infectious disease, or evidence of active or latent tuberculosis infection.
6. Clinical symptoms, signs, laboratory tests, or X-rays suggest active or latent tuberculosis Tuberculosis infected persons;
7. Those who have participated in any clinical study for any drug or medical device within 3 months before screening
8. Those who have received live attenuated vaccine within 12 weeks prior to screening or plan to receive live attenuated vaccine during the trial.
9. Blood donation or blood loss ≥ 400 mL within 8 weeks prior to screening, or receiving blood transfusion within 8 weeks;
10. Venous blood collection difficulties or physical conditions can not withstand blood collection;
11. Had used other drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines and dietary supplements) in the 2 weeks before screening;
12. Current or past alcoholics (drinking more than 14 standard units per week) 1 Standard unit containing 14g of alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); Or who cannot abstain from alcohol during the trial;
13. The average daily smoking amount in the 3 months before the test was ≥ 10 cigarettes; Or cannot stop using any tobacco products during the trial
14. History or evidence of ongoing alcohol or drug abuse, within the last six months before Baseline.
15. Female and male subjects who are fertile (defined as having the physical conditions necessary to become pregnant) who plan to become pregnant or donate sperm/egg within 20 weeks of using the study drug (greater than 5 half-lives) or who do not wish to use contraception; Female subjects who are fertile but have not used contraception in the 30 days prior to randomization;
16. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
17. Subjects judged by the investigator as unsuitable for participating in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-12-24 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
After a single subcutaneous injection of SHR-1314, assess injection site pain by VISUAL ANALOG SCALE at immediately after administration, 1 h, 48 h, Day 5 and Day 8, the results ranger from 0 to 10 cm, with higher scores indicating greater pain | Day 1 to Day 8 after each administration
After a single subcutaneous injection of SHR-1314, the incidence rate of injection site reaction at 1 h, 48 h, Day 5 and Day 8 | Day 1 to Day 8 after each administration

SECONDARY OUTCOMES:
After a single subcutaneous injection of SHR-1314, the PK parameters of plasma SHR-1314: Time to maximum concentration (Tmax) | Day 1 to Day 28
After a single subcutaneous injection of SHR-1314, the PK parameters of plasma SHR-1314: Area Under the Concentration versus time curve (AUC0-t) | Day 1 to Day 28
After a single subcutaneous injection of SHR-1314, the PK parameters of plasma SHR-1314: Maximum Concentration (Cmax) | Day 1 to Day 28
Safety indicators: The rate of adverse events (AE, including Injection site reactions), serious adverse events (SAE) | Screening period up to Day 43
Immunogenicity indicators: The rate of anti-SHR-1314 antibodies | Start of treatment up to Day 43

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dong Y, Gao X, Feng S, Lin L, Shen K, Hu W. Safety, pharmacokinetics, and bioequivalence of vunakizumab injection, a specific dermatitis drug, in healthy Chinese volunteers: an open-label, randomized, two-stage, two-sequence cross-over study. Expert Opin Drug Metab Toxicol. 2025 Sep;21(9):1117-1123. doi: 10.1080/17425255.2025.2558829. Epub 2025 Sep 15. PMID 40947125